CLINICAL TRIAL: NCT02845557
Title: Glucose Homeostasis, Incretin Effect and Cardiovascular Risk Burden in T2DM in the Youth- a Study of the Malaysian Population
Brief Title: Glucose Homeostasis and Incretin Effect T2DM in the Youth- a Study of the Malaysian Population
Status: Completed | Type: Observational
Sponsor: RCSI & UCD Malaysia Campus (Other)
Collaborators: Sarawak General Hospital (Other); Putrajaya Hospital, Malaysia (Unknown); Penang Hospital, Malaysia (Other Government); Institute of Neuroscience, Padova, Italy (Unknown); University of Copenhagen (Other); Institute for Medical Research, Malaysia (Unknown); Seberang Jaya Clinical Research Centre (Other Government)
Responsible Party: Principal Investigator, Toh-Peng Yeow, Associate Professor Dr., RCSI & UCD Malaysia Campus
Other Study IDs: NMRR-12-1042-13254
Record Dates: First submitted 2016-07-11; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Youth; Type 2 Diabetes; glucose homeostasis; incretin effect
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control subjects without diabetes: (i) 2-hour 75g OGTT with sampling of glucose, insulin, C-peptide and GLP-1 hormone, with sampling at fasting (time zero) and 30, 60, 90, 120 min after the glucose load.
  (ii) 1-hour IVGTT, with sampling at time 10 and 1 min, after which glucose (300 mg/kg body weight) infused in a contralateral vein within 30 s, starting at time zero. Blood further sampled for glucose, insulin and C-Peptide with sampling schedule: 3, 5, 6, 8, 10, 15, 20, 25,30 ,40 ,50 ,60 min;
  (iii) computed tomography scan, (CT) for abdominal subcutaneous and visceral fat quantification.
  Interventions: Other: OGTT and IVGTT tests
- Subjects with type 2 diabetes: (i) 2-hour 75g OGTT with sampling of glucose, insulin, C-peptide and GLP-1 hormone, with sampling at fasting (time zero) and 30, 60, 90, 120 min after the glucose load.
  (ii) 1-hour IVGTT, with sampling at time 10 and 1 min, after which glucose (300 mg/kg body weight) infused in a contralateral vein within 30 s, starting at time zero. Blood further sampled for glucose, insulin and C-Peptide with sampling schedule: 3, 5, 6, 8, 10, 15, 20, 25,30 ,40 ,50 ,60 min;
  (iii) computed tomography scan, (CT) for abdominal subcutaneous and visceral fat quantification.
  Interventions: Other: OGTT and IVGTT tests

INTERVENTIONS:
Other: OGTT and IVGTT tests

SUMMARY:
Early onset type 2 diabetes mellitus among adolescents/youth (YT2DM) is a rising phenomenon. The pathophysiology has been studied primarily on non-Asian populations while literature on incretin effect is scarce. The investigators evaluated insulin sensitivity, beta-cell function, incretin hormones and their effect in YT2DM from a multiethnic Malaysian population. The characterization of this population may enable us to better tailor their antidiabetic care.

DETAILED DESCRIPTION:
* The prevalence of Type 2 Diabetes Mellitus (T2DM) in the youth is increasing. Until 10 years ago in USA, T2DM accounted for less than 3% of all cases of new onset diabetes in adolescents. More recent data suggest up to 45% of cases are attributed to it.
* The prevalence of Diabetes Mellitus in Malaysia has risen from 11.6% to 15.2% over the last 5 years according to the National Health and Morbidity Survey in 2011. Among the population age 20-24 years old, the prevalence of diabetes has risen also from 2.0% to 4.9%. Of greater concern still is 90% of these young diabetes were previously undiagnosed, thus raising the possibility that these were predominantly T2DM. The report from the Malaysian DiCare registry (2006-2007) shows that T2DM accounted for 17.6% of diabetes in adolescents. In a more recent audit of diabetes clinic in Penang General Hospital in 2012, 56.7% of patients under age of 20 have clinical T2DM (data yet unpublished). The marked difference in proportion of young T2DM in both audits may be contributed by possible under-reporting in the first audit but raise the possibility also of rising incidence of young T2DM in Malaysia.
* This rising prevalence of T2DM in the youth has significant public health challenge. Studies in young adults have suggested that the development and progression of clinical complications might be especially rapid when the onset of T2DM is early. This, coupled with longer lifetime exposure to diabetes, raises the possibility of a serious public health challenge in the next few decades. Detailed understanding of the pathophysiology and complications burden among this population is therefore crucial to the development of appropriate management plan.
* Studies of youth onset T2DM suggest that it is driven by a combination of insulin resistance and beta cell dysfunction, and hyperglycemia does not develop until the beta cell fails to compensate appropriately to the peripheral insulin resistance state. However, these studies are predominantly done among the western populations and mainly in the Black and Hispanic ethnic groups. There are reasons to believe that pathophysiology may be different in different populations. The ability of the beta cell to secrete sufficient insulin to adequately respond to the peripheral insulin resistance state is influenced by genetic and environmental factors. Degree of insulin resistance appears to vary among different population studies. There is currently a paucity of literature with regards to pathophysiology underpinning T2DM among the Malaysian youth.
* The knowledge that incretin effect is severely reduced in patients with adult onset T2DM has been used to good pharmacotherapeutic effect in the patients. However, the incretin effect is less well studied among T2DM in the youth and understanding in this area will be helpful in guiding the use of incretin hormone for treatment of youth onset T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Youth with T2DM diagnosed at less than 25 years old
* The diagnosis of T2DM established based on the American Diabetes Association criteria for diabetes and absence of GAD antibodies and islet cell antibodies (ICAs).

Exclusion Criteria:

* Subjects with Type 1 Diabetes or secondary Diabetes
* Patients on medication that may impair glucose metabolism (e.g., steroids)
* Pregnancy

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 30 youths with type 2 diabetes with 18 gender- and age-matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Quantitative Insulin Sensitivity Check Index (QUICKI) | 1 year
  This is a cross sectional study where the outcome was measured whenever the test was conducted.
Oral Glucose Insulin Sensitivity Index (OGIS) | 1 year
  This is a cross sectional study where the outcome was measured whenever the test was conducted.
Early phase insulin response during OGTT was calculated for the first 30 minutes | 1 year
  This is a cross sectional study where the outcome was measured whenever the test was conducted.
Area under the curve for incretin hormone | 1 year
  This is a cross sectional study where the outcome was measured whenever the test was conducted.

SECONDARY OUTCOMES:
Incretin effect | 1 year
  It is estimated by relating the differences in beta cell responses from C peptide between stimulation with oral and intravenous glucose. The incretin effect is estimated by the formula 100 ×(BCOG BCIV)/BCOG).

CONTACTS AND LOCATIONS:
Locations (1):
- Penang Medical College, George Town, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wadwa RP, Urbina EM, Anderson AM, Hamman RF, Dolan LM, Rodriguez BL, Daniels SR, Dabelea D; SEARCH Study Group. Measures of arterial stiffness in youth with type 1 and type 2 diabetes: the SEARCH for diabetes in youth study. Diabetes Care. 2010 Apr;33(4):881-6. doi: 10.2337/dc09-0747. Epub 2010 Jan 12. PMID 20067960
- [Background] Malloy J, Capparelli E, Gottschalk M, Guan X, Kothare P, Fineman M. Pharmacology and tolerability of a single dose of exenatide in adolescent patients with type 2 diabetes mellitus being treated with metformin: a randomized, placebo-controlled, single-blind, dose-escalation, crossover study. Clin Ther. 2009 Apr;31(4):806-15. doi: 10.1016/j.clinthera.2009.04.005. PMID 19446153
- [Result] Rosenbloom AL, Silverstein JH, Amemiya S, Zeitler P, Klingensmith GJ. Type 2 diabetes in children and adolescents. Pediatr Diabetes. 2009 Sep;10 Suppl 12:17-32. doi: 10.1111/j.1399-5448.2009.00584.x. No abstract available. PMID 19754615
- [Result] D'Adamo E, Caprio S. Type 2 diabetes in youth: epidemiology and pathophysiology. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S161-5. doi: 10.2337/dc11-s212. No abstract available. PMID 21525449
- [Result] Pinhas-Hamiel O, Zeitler P. Acute and chronic complications of type 2 diabetes mellitus in children and adolescents. Lancet. 2007 May 26;369(9575):1823-1831. doi: 10.1016/S0140-6736(07)60821-6. PMID 17531891
- [Result] Maahs DM, Snively BM, Bell RA, Dolan L, Hirsch I, Imperatore G, Linder B, Marcovina SM, Mayer-Davis EJ, Pettitt DJ, Rodriguez BL, Dabelea D. Higher prevalence of elevated albumin excretion in youth with type 2 than type 1 diabetes: the SEARCH for Diabetes in Youth study. Diabetes Care. 2007 Oct;30(10):2593-8. doi: 10.2337/dc07-0450. Epub 2007 Jul 13. PMID 17630264
- [Result] Hillier TA, Pedula KL. Complications in young adults with early-onset type 2 diabetes: losing the relative protection of youth. Diabetes Care. 2003 Nov;26(11):2999-3005. doi: 10.2337/diacare.26.11.2999. PMID 14578230
- [Result] Gungor N, Bacha F, Saad R, Janosky J, Arslanian S. Youth type 2 diabetes: insulin resistance, beta-cell failure, or both? Diabetes Care. 2005 Mar;28(3):638-44. doi: 10.2337/diacare.28.3.638. PMID 15735201
- [Result] Umpaichitra V, Bastian W, Taha D, Banerji MA, AvRuskin TW, Castells S. C-peptide and glucagon profiles in minority children with type 2 diabetes mellitus. J Clin Endocrinol Metab. 2001 Apr;86(4):1605-9. doi: 10.1210/jcem.86.4.7415. PMID 11297591
- [Result] Kobayashi K, Amemiya S, Higashida K, Ishihara T, Sawanobori E, Kobayashi K, Mochizuki M, Kikuchi N, Tokuyama K, Nakazawa S. Pathogenic factors of glucose intolerance in obese Japanese adolescents with type 2 diabetes. Metabolism. 2000 Feb;49(2):186-91. doi: 10.1016/s0026-0495(00)91221-6. PMID 10690942
- [Result] Musso G, Gambino R, Pacini G, De Michieli F, Cassader M. Prolonged saturated fat-induced, glucose-dependent insulinotropic polypeptide elevation is associated with adipokine imbalance and liver injury in nonalcoholic steatohepatitis: dysregulated enteroadipocyte axis as a novel feature of fatty liver. Am J Clin Nutr. 2009 Feb;89(2):558-67. doi: 10.3945/ajcn.2008.26720. Epub 2009 Jan 13. PMID 19141695
- [Result] Pacini G, Tura A, Winhofer Y, Kautzky-Willer A. Incretin Effect in Women with Former Gestational Diabetes within a Short Period after Delivery. Int J Endocrinol. 2012;2012:247392. doi: 10.1155/2012/247392. Epub 2012 Apr 19. PMID 22577378
- [Result] Danadian K, Balasekaran G, Lewy V, Meza MP, Robertson R, Arslanian SA. Insulin sensitivity in African-American children with and without family history of type 2 diabetes. Diabetes Care. 1999 Aug;22(8):1325-9. doi: 10.2337/diacare.22.8.1325. PMID 10480778
- [Result] Kvist H, Chowdhury B, Grangard U, Tylen U, Sjostrom L. Total and visceral adipose-tissue volumes derived from measurements with computed tomography in adult men and women: predictive equations. Am J Clin Nutr. 1988 Dec;48(6):1351-61. doi: 10.1093/ajcn/48.6.1351. PMID 3202084
- [Result] McQuaid S, O'Gorman DJ, Yousif O, Yeow TP, Rahman Y, Gasparro D, Pacini G, Nolan JJ. Early-onset insulin-resistant diabetes in obese Caucasians has features of typical type 2 diabetes, but 3 decades earlier. Diabetes Care. 2005 May;28(5):1216-8. doi: 10.2337/diacare.28.5.1216. No abstract available. PMID 15855595
- [Result] Pacini G, Tonolo G, Sambataro M, Maioli M, Ciccarese M, Brocco E, Avogaro A, Nosadini R. Insulin sensitivity and glucose effectiveness: minimal model analysis of regular and insulin-modified FSIGT. Am J Physiol. 1998 Apr;274(4):E592-9. doi: 10.1152/ajpendo.1998.274.4.E592. PMID 9575818
- [Result] Ahren B, Pacini G. Importance of quantifying insulin secretion in relation to insulin sensitivity to accurately assess beta cell function in clinical studies. Eur J Endocrinol. 2004 Feb;150(2):97-104. doi: 10.1530/eje.0.1500097. PMID 14763905
- [Result] Knop FK, Aaboe K, Vilsboll T, Volund A, Holst JJ, Krarup T, Madsbad S. Impaired incretin effect and fasting hyperglucagonaemia characterizing type 2 diabetic subjects are early signs of dysmetabolism in obesity. Diabetes Obes Metab. 2012 Jun;14(6):500-10. doi: 10.1111/j.1463-1326.2011.01549.x. Epub 2012 Jan 17. PMID 22171657
- [Result] Pacini G, Mari A. Methods for clinical assessment of insulin sensitivity and beta-cell function. Best Pract Res Clin Endocrinol Metab. 2003 Sep;17(3):305-22. doi: 10.1016/s1521-690x(03)00042-3. PMID 12962688
- [Result] Bloomgarden ZT. Type 2 diabetes in the young: the evolving epidemic. Diabetes Care. 2004 Apr;27(4):998-1010. doi: 10.2337/diacare.27.4.998. No abstract available. PMID 15047665
- [Result] Svec F, Nastasi K, Hilton C, Bao W, Srinivasan SR, Berenson GS. Black-white contrasts in insulin levels during pubertal development. The Bogalusa Heart Study. Diabetes. 1992 Mar;41(3):313-7. doi: 10.2337/diab.41.3.313. PMID 1551490
- [Result] Yokoyama H, Okudaira M, Otani T, Takaike H, Miura J, Saeki A, Uchigata Y, Omori Y. Existence of early-onset NIDDM Japanese demonstrating severe diabetic complications. Diabetes Care. 1997 May;20(5):844-7. doi: 10.2337/diacare.20.5.844. PMID 9135953
- [Result] TODAY Study Group; Zeitler P, Hirst K, Pyle L, Linder B, Copeland K, Arslanian S, Cuttler L, Nathan DM, Tollefsen S, Wilfley D, Kaufman F. A clinical trial to maintain glycemic control in youth with type 2 diabetes. N Engl J Med. 2012 Jun 14;366(24):2247-56. doi: 10.1056/NEJMoa1109333. Epub 2012 Apr 29. PMID 22540912